CLINICAL TRIAL: NCT03663075
Title: The Effect of Group and Individual Counseling on Mental Health, Quality of Life and Sick Leave in 45-60 Year Old Women With Stress Related Symptoms - A Randomized Controlled Trial
Brief Title: Effect of Group Education and Individual Counselling on Mental Health and Quality of Life in 45-60 Year Old Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1219-6542
Record Dates: First submitted 2018-08-29; First posted 2018-09-10 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2020-11

CONDITIONS: Women's Health; Quality of Life; Mental Health; Menopause; Primary Health Care; Sick Leave
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Two factor design evaluating two separate treatment modalities
Masking Description: This study evaluated the effect of groups sessions or individual support. This is not a pill so it is impossible to mask participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): This group will receive the intervention Group information (GI).
  Interventions: Behavioral: Group information (GI)
- Group 2 (Experimental): This group will receive the intervention Group information (GI) followed by Structured person-centered support (PCS)
  Interventions: Behavioral: Group information (GI); Behavioral: Structured person-centered support (PCS)
- Group 3 (Experimental): This group will receive the intervention Structured person-centered support (PCS)
  Interventions: Behavioral: Structured person-centered support (PCS)
- Group 4 (No Intervention): This is a control group.

INTERVENTIONS:
Behavioral: Group information (GI) — The group education consists of four information sessions discussing myths and myths around menopause, physiology, local estrogen deficiency symptoms, women's cardiovascular health, stress-related ill health, mental health, relationships, sexuality, lust and possible treatment options. In addition, conversations about insight into obstacles and resources, coping strategies and behavioral changes will be included.
  Arms: Group 1; Group 2
Behavioral: Structured person-centered support (PCS) — The individually structured person-centered support comprises of five meetings consisting of dialogue on symptoms of stress-related ill health, physiology and coping strategies.
  Arms: Group 2; Group 3

SUMMARY:
Background:

Stress-related ill health is today the most common cause of long-term sick leave in women in the middle of life and a common cause of visits to primary health care.

Objective:

To implement and investigate the effect of education in group and/or individually held in primary health care clinics embracing aspects of mental health, quality of life, sick leave and the needs women aged 45-60 with stress-related symptoms have.

Method The study is a randomized controlled trial with a two-factor design. The study evaluates both group information (GI) and structured person-centered support (PCS) and possible interaction effects between these two treatment modalities. The group education consists of four information sessions discussing myths around menopause, physiology, local estrogen deficiency symptoms, women's cardiovascular health, stress-related ill health, mental health, relationships, sexuality, lust and possible treatment options. In addition, conversations about insight into obstacles and resources, coping strategies and behavioral changes will be included. The individually structured person-centered support comprises of five meetings consisting of dialogue on symptoms of stress-related ill health, physiology and coping strategies. Participants will be block randomized into four groups; GI, PCS, GI+PCS or control.

Expected result Implementation of group and individual support calls is expected to improve health for women seeking primary care care. The results are expected to increase the knowledge of how women's health is affected by short-term care in primary care through reduced sick leave days, reduced care needs, return to work and increased quality of life. The result may improve existing primary care routines for women, and if needed, for a more individualized care contact and support.

DETAILED DESCRIPTION:
Background:

Stress-related ill health is today the most common cause of long-term sick leave in women in the middle of life and a common cause of visits to primary health care. Women seem to suffer more than men in the same age group. Few evidence based treatment options exist and none of them has a proven effect on return to work.

Objective:

To implement and investigate the effect of education in group and/or individually held in primary health care clinics embracing aspects of mental health, quality of life, sick leave and the needs women aged 45-60 with stress-related symptoms have.

Method The study is a randomized controlled trial with a two-factor design. The study evaluates both group information (GI) and structured person-centered support (PCS) and possible interaction effects between these two treatment modalities. The group education consists of four information sessions discussing myths around menopause, physiology, local estrogen deficiency symptoms, women's cardiovascular health, stress-related ill health, mental health, relationships, sexuality, lust and possible treatment options. In addition, conversations about insight into obstacles and resources, coping strategies and behavioral changes will be included. The individually structured person-centered support comprises of five meetings consisting of dialogue on symptoms of stress-related ill health, physiology and coping strategies. Participants will be block randomized into four groups; GI, PCS, GI+PCS or control.

Expected result Implementation of group and individual support calls is expected to improve health for women seeking primary care care. The results are expected to increase the knowledge of how women's health is affected by short-term care in primary care through reduced sick leave days, reduced care needs, return to work and increased quality of life. The result may improve existing primary care routines for women, and if needed, for a more individualized care contact and support.

ELIGIBILITY:
Inclusion Criteria:

* The woman has at least one possible stress related problem such as depression, anxiety, gastrointestinal disturbance, unexplained muscular pain or cardiovascular illness such as hypertension or coronary heart disease.
* The woman have not been on sick leave for more than 30 days during the preceding 60 days.
* The woman can easily understand and communicate freely in the Swedish language.
* The woman does not have severe mental illness such as schizophrenia, other psychosis or known neuropsychiatric disorder. The woman is not in terminal palliative care.
* The woman does not have severe depression (MADRS scores >20 or express suicidal ideation)

Exclusion Criteria:

* The woman do not wish to continue participation

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study specifically aim to study women in the age 45-60 years attending primary health care for stress related symptoms.
Enrollment: 370 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Short term effect of group education (GI) on change in quality of life | Change from baseline to six months after completed intervention
  What is the effect of group education (GI) on quality of life (measured by change in scores in SF36 from baseline to 6 months after completed intervention)

SECONDARY OUTCOMES:
Short term effect of Structured person-centered support (PCS) on change in days on sick leave | Change from baseline to six months after completed intervention
  What is the effect of Structured person-centered support (PCS) on change in number of days on sick leave. (At baseline the number of days on sick leave up until present time is stated by women currently being on sick leave. At the 6 month follow the same information is retrieved is retrieved. The change is the difference between these measurements.)
Short term effect of Structured person-centered support (PCS) on change in depressive mood | Change from baseline to six months after completed intervention
  What is the effect of Structured person-centered support (PCS) on depressive mood (measured by change in scores in MADRS from baseline to 6 months after completed intervention)
Short term effect of Structured person-centered support (PCS) on change in quality of life | Change from baseline to six months after completed intervention
  What is the effect of Structured person-centered support (PCS) on quality of life (measured by change in scores in SF36 from baseline to 6 months after completed intervention)
Short term effect of Structured person-centered support (PCS) on stress levels | Change from baseline to six months after completed intervention
  What is the effect of Structured person-centered support (PCS) on stress levels (measured by change in scores in PSS-14 from baseline to 6 months after completed intervention)
Short term effect of group education (GI) on change in days on sick leave | Change from baseline to six months after completed intervention
  What is the effect of group education (GI) on change in number of days on sick leave. (At baseline the number of days on sick leave up until present time is stated by women currently being on sick leave. At the 6 month follow the same information is retrieved is retrieved. The change is the difference between these measurements.)
Short term effect of group education (GI) on change in depressive mood | Change from baseline to six months after completed intervention
  What is the effect of group education (GI) on depressive mood (measured by change in scores in MADRS from baseline to 6 months after completed intervention)
Short term effect of group education (GI) on stress levels | Change from baseline to six months after completed intervention
  What is the effect of group education (GI) on stress levels (measured by change in scores in PSS-14 from baseline to 6 months after completed intervention).
Long term effect of Structured person-centered support (PCS) on change in days on sick leave | Change from baseline to 12 months after completed intervention
  What is the effect of Structured person-centered support (PCS) on change in number of days on sick leave. (At baseline the number of days on sick leave up until present time is stated by women currently being on sick leave. At the 12 month follow the same information is retrieved is retrieved. The change is the difference between these measurements.)
Long term effect of Structured person-centered support (PCS) on change in depressive mood | Change from baseline to 12 months after completed intervention
  What is the effect of Structured person-centered support (PCS) on depressive mood (measured by change in scores in MADRS from baseline to 12 months after completed intervention)
Long term effect of Structured person-centered support (PCS) on change in quality of life | Change from baseline to 12 months after completed intervention
  What is the effect of Structured person-centered support (PCS) on quality of life (measured by change in scores in SF36 from baseline to 12 months after completed intervention)
Long term effect of Structured person-centered support (PCS) on stress levels | Change from baseline to 12 months after completed intervention
  What is the effect of Structured person-centered support (PCS) on stress levels (measured by change in scores in PSS-14 from baseline to 12 months after completed intervention)
Long term effect of group education (GI) on change in days on sick leave | Change from baseline to 12 months after completed intervention
  What is the effect of group education (GI) on change in number of days on sick leave. (At baseline the number of days on sick leave up until present time is stated by women currently being on sick leave. At the 12 month follow the same information is retrieved is retrieved. The change is the difference between these measurements.)
Long term effect of group education (GI) on change in depressive mood | Change from baseline to 12 months after completed intervention
  What is the effect of group education (GI) on depressive mood (measured by change in scores in MADRS from baseline to 12 months after completed intervention)
Long term effect of group education (GI) on change in quality of life | Change from baseline to 12 months after completed intervention
  What is the effect of group education (GI) on quality of life (measured by change in scores in SF36 from baseline to 12 months after completed intervention)
Long term effect of group education (GI) on stress levels | Change from baseline to 12 months after completed intervention
  What is the effect of group education (GI) on stress levels (measured by change in scores in PSS-14 from baseline to 12 months after completed intervention).
Short term effect of group education (GI) on levels of anxiety | Change from baseline to 6 months after completed intervention
  What is the effect of group education (GI) on stress levels (measured by change in scores in HAD from baseline to 6 months after completed intervention).
Long term effect of group education (GI) on levels of anxiety | Change from baseline to 12 months after completed intervention
  What is the effect of group education (GI) on stress levels (measured by change in scores in HAD from baseline to 12 months after completed intervention).
Short term effect of Structured person-centered support (PCS) on levels of anxiety | Change from baseline to 6 months after completed intervention
  What is the effect of Structured person-centered support (PCS) on stress levels (measured by change in scores in HAD from baseline to 6 months after completed intervention).
Long term effect of Structured person-centered support (PCS) on levels of anxiety | Change from baseline to 12 months after completed intervention
  What is the effect of Structured person-centered support (PCS) on stress levels (measured by change in scores in HAD from baseline to 12 months after completed intervention).
Short term effect of Structured person-centered support (PCS) on visits to primary health care | Change from baseline to 6 months after completed intervention
  What is the effect of Structured person-centered support (PCS) on visits to primary health care (women are asked at baseline if they had to visit the primary health care center during the preceding two months. The same question is asked at 6 months. The measurement is the change in proportion of women who visited the primary health care center).
Long term effect of Structured person-centered support (PCS) on visits to primary health care | Change from baseline to 12 months after completed intervention
  What is the effect of Structured person-centered support (PCS) on visits to primary health care (women are asked at baseline if they had to visit the primary health care center during the preceding two months. The same question is asked at 12 months. The measurement is the change in proportion of women who visited the primary health care center).
Short term effect of group education (GI) on visits to primary health care | Change from baseline to 6 months after completed intervention
  What is the effect of group education (GI) on visits to primary health care (women are asked at baseline if they had to visit the primary health care center during the preceding two months. The same question is asked at 6 months. The measurement is the change in proportion of women who visited the primary health care center).
Long term effect of group education (GI) on visits to primary health care | Change from baseline to 12 months after completed intervention
  What is the effect of group education (GI) on visits to primary health care (women are asked at baseline if they had to visit the primary health care center during the preceding two months. The same question is asked at 12 months. The measurement is the change in proportion of women who visited the primary health care center).

CONTACTS AND LOCATIONS:
Overall Officials: Lena Rindner, Principal Investigator — Vastra Gotaland region, Sweden
Locations (1):
- Research and Development Unit, Borås, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
The descriptive data provided will be summary data for each group. The investigators will not show data from single participants.

REFERENCES:
- [Result] Rindner L, Nordeman L, Stromme G, Hange D, Gunnarsson R, Rembeck G. Effect of group education and person-centered support in primary health care on mental health and quality of life in women aged 45-60 years with symptoms commonly associated with stress: a randomized controlled trial. BMC Womens Health. 2023 Mar 24;23(1):128. doi: 10.1186/s12905-023-02221-6. PMID 36964526

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT03663075/Prot_SAP_000.pdf